CLINICAL TRIAL: NCT02610517
Title: Integration of Evidence-based Alcohol Interventions Into HIV Care (ARCH-IRA) (Phases 1- Provider Training and 2- Patient Intervention)
Brief Title: ARCH Research Protocol for Provider Alcohol Pharmacotherapy Training and Assessment
Acronym: ARCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Washington (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Michael Saag, MD, Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: F121009007
Record Dates: First submitted 2015-08-29; First posted 2015-11-20 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: HIV; Alcoholism
Keywords: Hazardous alcohol use; Computer based intervention (CBI); Pharmacotherapy
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Provider Training (Other): Training providers to offer alcohol pharmacotherapy to at-risk drinkers interested in quitting or reducing their drinking as part of overall HIV care could be an important strategy to reduce hazardous alcohol use in this medically-ill population.
  Interventions: Behavioral: Provider Training
- Patient Intervention (Other): Determine the effectiveness of a computer-delivered brief intervention (CBI) for reducing hazardous drinking in the HIV clinical care setting at two intervention clinics: University of Alabama at Birmingham (UAB) and the University of Washington (UW).
  Interventions: Behavioral: Patient Intervention

INTERVENTIONS:
Behavioral: Provider Training — All providers will receive an online survey about alcohol pharmacotherapy, and an on-site training on alcohol pharmacotherapy will be offered at UAB and UW. The training will cover the most commonly prescribed alcohol pharmacotherapy. Some medications (ex: Zofran) have been used clinically for alcohol pharmacotherapy but have not yet received FDA approval for this indication. Research has shown these medications are beneficial as alcohol pharmacotherapy and are more frequently used by doctors due to the more favorable side effects. Providers in this study will use their clinical judgment in prescribing alcohol medications per their normal standard of care and using any new information gained from the alcohol pharmacotherapy training.
  Arms: Provider Training
Behavioral: Patient Intervention — Eligible participants will be screened using the Audit and Mini instruments that are routinely asked during regular clinic visits. Once a participant consents, they will be shown 2 computerized brief interventions (CBIs) - one after enrollment (visit 1) and one 3-6 months after enrollment (visit 2). Participants will interact with the touch-screen computer via Peedy the Parrot, a three dimensional animated character. The intervention emphasizes personal responsibility for change, uses empathy as a counseling style, and enhances self-efficacy. At the end of both visits, patients will complete a patient satisfaction survey with questions related to ease of use of CBI and satisfaction with program content. Providers will have the opportunity to prescribe pharmacotherapy at visit 1 and 2.
  Arms: Patient Intervention

SUMMARY:
Phase 1: To train providers to offer alcohol pharmacotherapy to at-risk drinkers interested in quitting or reducing their drinking as part of overall HIV care. Phase 2: To determine the effectiveness of a computer-delivered brief intervention (CBI) for reducing hazardous drinking in the HIV clinical care setting.

DETAILED DESCRIPTION:
This study is divided into 2 phases: provider training (Phase 1) and patient level intervention (Phase 2). Phase 1, provider training, is managed through an administrative grant at Johns Hopkins. Providers will be notified of the research project locally but all training and assessments will be through Johns Hopkins.

Phase 1:

Training providers to offer alcohol pharmacotherapy (APT) to at-risk drinkers interested in quitting or reducing their drinking as part of overall HIV care could be an important strategy to reduce hazardous alcohol use in this medically-ill population. However, it is unknown how Infectious Disease providers will feel about treating alcohol use disorders within HIV clinics. Further it is uncertain the specific provider and clinic barriers to implementing this type of program in a primary care setting. A web-based alcohol pharmacotherapy provider training will be provided across the Center for AIDS Research (CFAR) Network of Integrated Clinical Systems (CNICS), a national network of 8 clinical cohorts. At the two intervention sites (University of Alabama at Birmingham and the University of Washington), providers will receive an on-site training in addition to the web-based training on alcohol pharmacotherapy administered at all 8 sites.

The following are the specific aims of this project:

Aim 1: To evaluate provider attitudes before and after alcohol pharmacotherapy training.

Aim 2: To determine barriers and facilitators to alcohol treatment implementation in HIV specialty clinics.

Phase 2:

Determine the effectiveness of computer-delivered brief interventions (CBI) for reducing hazardous drinking in the HIV clinical care setting at two intervention clinics: University of Alabama at Birmingham (UAB) and the University of Washington (UW). The combination of CBI plus alcohol pharmacotherapy (APT) provider training (Phase 1) will be piloted in two clinics in the Center for AIDS Research (CFAR) Network of Integrated Clinical Systems (CNICS), a national network of 8 clinical cohorts. Across all 8 CNICS sites, all patients will be screened for hazardous or binge drinking using the AUDIT (Alcohol Use Disorders Identification Test) and MINI (Mini-International Neuropsychiatric Interview) instruments. At UAB and UW, patients who screen eligible (self-report of hazardous or binge drinking using the AUDIT and MINI instruments) will be approached for participation. The data collected through this protocol will be used to compare Standard of Care as noted in Aim 2 below. Standard of Care at UAB includes potential referral to an in-house substance abuse program or an outside agency, both of which are based on the provider's discretion. Providers have the option of offering alcohol pharmacotherapy but this has not been used to date routinely.

Specific aims of this proposal are:

Aim 1: Develop a tailored CBI intervention that addresses alcohol risks specific to HIV-infected patients.

Aim 2: Compare the effectiveness of CBI + APT versus standard care for reducing alcohol use among hazardous drinking HIV infected individuals.

Aim 3: Determine patient-level predictors of CBI and APT engagement and effectiveness.

Aim 4: Determine the facilitators and barriers to successful integration and implementation of these interventions into HIV clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years or older
* Receiving HIV care at The UAB 1917 Clinic
* Hazardous drinkers as defined by an at-risk alcohol use score on the alcohol related, self-report data collected through the CNICS PRO.
* English speaking
* Willing to participate and provide informed consent

Exclusion Criteria:

* Pregnant or nursing women will be referred to social work for more intensive intervention per standard of care.
* Cognitive impairment such as they cannot provide informed consent
* Non-English speaker
* A visibly intoxicated person will be deferred for consent by the research assistant but will remain eligible for the study
* Patients who previously declined to participate in the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Drinks per week | up to 1 year after enrollment
  The Alcohol Use Disorders Identification Test (AUDIT) instrument will be used to assess drinks per week. This is a self-reported instrument.
Binge drinking episodes | up to 1 year after enrollment
  The Mini-International Neuropsychiatric Interview (MINI) instrument will be used to assess binge drinking episodes. This is a self-reported instrument.

SECONDARY OUTCOMES:
Number of participants that initiate/request alcohol pharmacotherapy | at enrollment and after visit 2 (3 - 6 months after enrollment)
  Prescription of alcohol pharmacotherapy - number of participants obtaining a prescription at enrollment and/or after visit 2.
Number of participants that complete a CNICS Patient Reported Outcome (PRO) | every 3 - 6 months after enrollment and at 12 months after enrollment
  The CNICS PRO is a patient self-reported questionnaire that is asked every 3 - 6 months during a regular clinic visit. The instruments that are used include:
  Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST); Adult AIDS Clinical Trials Group (AACTG) Adherence; HIV Risk Behaviors; Quality of Life (EuroQOL); Patient Health Questionnaire for Depression and Anxiety (PHQ-9 - Depression; PHQ-5 - Anxiety); Tobacco; Physical Activity
Number of participants that initiate antiretroviral therapy (ART) | every 3 - 6 months after enrollment and at 12 months after enrollment
  New prescription of ART if they previously were not on therapy
Mean number of participants that adhere to HIV clinic visits | for 1 year after enrollment
  Medical records data will be used to record the data
Number of subjects with HIV-RNA level (viral loads) < 20 copies/ml | 1 year post enrollment
  Virological suppression to < 20 copies/ml

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Saag, MD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Johns Hopkins University, Baltimore, Maryland
  - University of Washington, Seattle, Washington